CLINICAL TRIAL: NCT01997060
Title: Physiological Factors That Influence Maintenance of Lifestyle Changes and Weight Loss - a Longitudinal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Ubberup Folk High School (Other)
Responsible Party: Principal Investigator, Jørn Wulff Helge, Associate Professor, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UBBERUP2
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Obesity; Overweight
Keywords: Lifestyle intervention; Body weight; Body composition; Weight loss maintenance; Physical activity
MeSH Terms: conditions — Obesity; Overweight; Body Weight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intensive Lifestyle Intervention (Experimental): Intensive Lifestyle Intervention at Ubberup Folk High School for 10-14 weeks. Daily exercise for 1-3hrs. Calorie restriction (~-700KCal/day). Education within nutrition, exercise and healthy living in general.
  Interventions: Behavioral: Intensive Lifestyle Intervention

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention

SUMMARY:
In Denmark and the western world, there is an increasing prevalence of obesity probably due to a combination of inadequate daily physical activity and a high energy intake. One approach to achieve weight loss and change life style is to participate in an intensive supervised prolonged life style modification course. The immediate effect is often positive, but over time the overall effect is limited as the majority will not maintain weight loss and a changed life style.

The purpose of this study is therefore to characterize the physiological factors that determine/influence the capacity to maintain weight loss and a healthy lifestyle after a prolonged lifestyle intervention.

We have the following research questions:

1. Are there physiological traits and characteristics that mediate better adherence to lifestyle changes and weight loss?
2. Does the adaptation in muscle oxidative capacity after lifestyle intervention predict success in maintaining weight loss and lifestyle changes 3, 12 and 39 months after intervention?
3. How does gender and age influence the capacity to maintain the lifestyle induced adaptation in muscle and adipose tissue and maintaining weight loss?

The study design is a longitudinal intervention and will be based on a lifestyle intervention, as it is practiced in a real life setting at Ubberup folk high school.

ELIGIBILITY:
Inclusion Criteria:

* Participants at Ubberup Folk High School

Exclusion Criteria:

* Previous Gastric Bypass Surgery or Gastric Banding
* BMI<25

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Total body weight | Changes from baseline at 3, 6, 15 and 39 months

SECONDARY OUTCOMES:
Maximal fat oxidation during exercise | Changes from baseline at 3, 6, 15 and 39 months
  Respiratory Exchange Ratio (RER) is measured and maximal fat oxidation is calculated.
Anthropometry | Changes from baseline at 3, 6, 15 and 39 months
  Body composition measured by dual x-ray absorptiometry or bio-impedance, height, weight, waist circumference.
Maximal Oxygen Consumption | Changes from baseline at 3, 6, 15 and 39 months

OTHER OUTCOMES:
Adherence to physical activity | Changes from baseline at 3, 6, 15 and 39 months
  International Physical Activity Questionaire (IPAQ) to determine adherence to physical activity. Furthermore we will use diary and ActiHeart (accelerometer).
Adherence to healthy diet | Changes from baseline at 3, 6, 15 and 39 months
  Questionnaire (24hrs dietary recall) and diary to determine adherence to a healthy diet.
Mitochondria respiration and efficiency | Changes from baseline at 3, 6, 15 and 39 months
  Mitochondria respiration and efficiency is measured by Oreboros Oxygraph.
Blood and plasma substrates, hormones and metabolites | Changes from baseline at 3, 6, 15 and 39 months
  HbA1c, insulin, leptin, glucose, adiponectin, thyroid stimulating hormone (TSH), ghrelin
Muscle lipid composition | Changes from baseline at 3, 6, 15 and 39 months
  Muscle lipid composition will be analysed using a lipidomics approach.
Expression of muscle lipases | Changes from baseline at 3, 6, 15 and 39 months
  Western blot analysis will be applied to analyse expression of muscle lipases; hormone sensitive lipase (HSL), adipose triglyceride lipase (ATGL) and lipoprotein lipase (LPL) as well as muscle PAT proteins; PLIN 2 (ADRP), PLIN 3 (TIP47) and PLIN 5 (OXPAT)
Intramuscular lipid droplet content and size, glycogen content and ceramide content and location | Changes from baseline at 3, 6, 15 and 39 months
  Intramuscular lipid droplet content and size, glycogen content and ceramide content and location will be quantified by immunohistochemical staining of serial cryo-sections of muscle tissue samples that are visualized by confocal microscopy
Adipose tissue macrophage inflammation and cytokine production | Changes from baseline at 3, 6, 15 and 39 months
Motivation for lifestyle changes and sociological factors involved | Changes from baseline at 3, 6, 15 and 39 months
  Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jørn W Helge, PhD, Principal Investigator — University of Copenhagen, Department of Biomedical Sciences
Locations (1):
- University of Copenhagen, Department of Biomedical Sciences, Copenhagen, Denmark

REFERENCES:
- [Background] Karlsen TI, Sohagen M, Hjelmesaeth J. Predictors of weight loss after an intensive lifestyle intervention program in obese patients: a 1-year prospective cohort study. Health Qual Life Outcomes. 2013 Oct 3;11:165. doi: 10.1186/1477-7525-11-165. PMID 24090083
- [Background] McCormack SE, McCarthy MA, Harrington SG, Farilla L, Hrovat MI, Systrom DM, Thomas BJ, Torriani M, McInnis K, Grinspoon SK, Fleischman A. Effects of exercise and lifestyle modification on fitness, insulin resistance, skeletal muscle oxidative phosphorylation and intramyocellular lipid content in obese children and adolescents. Pediatr Obes. 2014 Aug;9(4):281-91. doi: 10.1111/j.2047-6310.2013.00180.x. Epub 2013 Jun 25. PMID 23801526
- [Background] Danielsen KK, Svendsen M, Maehlum S, Sundgot-Borgen J. Changes in body composition, cardiovascular disease risk factors, and eating behavior after an intensive lifestyle intervention with high volume of physical activity in severely obese subjects: a prospective clinical controlled trial. J Obes. 2013;2013:325464. doi: 10.1155/2013/325464. Epub 2013 Apr 22. PMID 23710347
- [Background] Bruun JM, Helge JW, Richelsen B, Stallknecht B. Diet and exercise reduce low-grade inflammation and macrophage infiltration in adipose tissue but not in skeletal muscle in severely obese subjects. Am J Physiol Endocrinol Metab. 2006 May;290(5):E961-7. doi: 10.1152/ajpendo.00506.2005. Epub 2005 Dec 13. PMID 16352667
- [Background] Pedersen JO, Zimmermann E, Stallknecht BM, Bruun JM, Kroustrup JP, Larsen JF, Helge JW. [Lifestyle intervention in the treatment of severe obesity]. Ugeskr Laeger. 2006 Jan 9;168(2):167-72. Danish. PMID 16403343
- [Background] Bruun JM, Stallknecht B, Helge JW, Richelsen B. Interleukin-18 in plasma and adipose tissue: effects of obesity, insulin resistance, and weight loss. Eur J Endocrinol. 2007 Oct;157(4):465-71. doi: 10.1530/EJE-07-0206. PMID 17893261
- [Background] Christiansen T, Bruun JM, Madsen EL, Richelsen B. Weight loss maintenance in severely obese adults after an intensive lifestyle intervention: 2- to 4-year follow-up. Obesity (Silver Spring). 2007 Feb;15(2):413-20. doi: 10.1038/oby.2007.530. PMID 17299115
- [Derived] Elsborg P, Elbe AM. Exercise-specific volition and motivation for weight loss maintenance following an intensive lifestyle intervention. Health Psychol. 2018 Aug;37(8):759-766. doi: 10.1037/hea0000636. PMID 30024231